CLINICAL TRIAL: NCT00504387
Title: Burning Mouth Disorder (BMD) - a Neuropathic Pain Disorder? An Investigation Using Qualitative and Quantitative Sensory Testing (QST)
Brief Title: Burning Mouth Disorder (BMD) - A Neuropathic Pain Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Markus R. Fussnegger (Other)
Collaborators: Deutsche Gesellschaft für Zahn-, Mund- und Kieferheilkunde e.V. (Unknown)
Responsible Party: Sponsor-Investigator, Markus R. Fussnegger, Assistent professor, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: EA4/036/06
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Burning Mouth Syndrome; Taste Disorder; Orofacial Pain
Keywords: Burning mouth disorder; Taste disorder; Quantitative sensory testing; Gustatory testing; Neuropathic orofacial pain; Oral burning
MeSH Terms: conditions — Burning Mouth Syndrome; Taste Disorders; Facial Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Patients: Patients with a primary burning mouth disorder Pain (VAS 0-10): 3<x<9 Patient understands and speaks german Age: >18 years
- B: Controls: Age and sex matched persons/patients who do not have any history of an oral burning sensation or a burning mouth disorder.

SUMMARY:
Oral burning can have a multitude of reasons. Recent neurophysiologic study results suggest that a primary burning mouth disorder (BMD) may be a peripheral and/or a central neuropathic disorder. The aim of this study is to first identify patients with a primary burning mouth disorder by excluding other possible causes for oral burning. By means of qualitative and quantitative sensory testing and a gustatory examination in the individual patient the investigators want to find out whether neurosensory differences exist between patients with a primary BMD and controls and whether gustatory and neurosensory deficits always coexist in BMD-patients.

DETAILED DESCRIPTION:
Oral burning can have many different etiologies. Secondary burning mouth disorders (BMD) due to systemic (i.e. diabetes, nutritional deficiencies, allergies), local (i.e. Candidiasis, Lichen planus) or functional factors (i.e. tongue parafunctional activities, mouth breathing) are usually fairly easy to identify and are treated by eliminating the respective cause. A primary BMD as a specific disease is a challenging disorder with regard to assessment and treatment for both, the patient and the dentist. The prevailing hypothesis of a predominantly psychological cause is questioned by recent research results. The typical burning sensation, the partly efficacy of medication that is usually used in chronic, neuropathic pains and recent neurophysiologic studies and finally the finding of a degeneration of epithelial nerve fibers in BMD patients give reason to assume a peripheral and/or central neuropathic etiology. That is, the transduction of nociceptive stimuli in the orofacial region and the transmission and modulation of the nociceptive input might be altered. The hypothesis of a disorder of the gustatory system assumes that gustatory input has an inhibitory influence on the trigeminal nociceptive system. A hypogeusia or ageusia, maybe caused by peripheral nerve degeneration that has been found in BMD patients would therefore lead to a decreased gustatory input which in turn gives way to a central disinhibition of trigeminal nociception, leading to a more painful perception in the oral region. The aim of this study is to first identify patients with a primary burning mouth disorder by excluding other possible causes for oral burning. By means of qualitative and thermal quantitative sensory testing and a gustatory examination in the individual patient we want to find out whether neurosensory differences exist between patients with a primary BMD and controls and whether gustatory and neurosensory deficits always coexist in BMD-patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary burning sensation of the tongue, lip or other oral structure
* Average pain intensity between 3 and 9 (VAS-Scale 0-10)
* Written, informed consent
* patient speaks German
* Age > 18 years old

Exclusion Criteria:

* Tumor
* HIV/AIDS
* Diabetes mellitus
* untreated hypothyroidism
* gastroesophageal reflux disease
* Sjögren's disease
* Salivary gland disease
* Vitamin B-, folic acid- and iron deficiency
* Medications causing hyposalivation
* Inflammatory, viral, bacterial, fungal, autoimmune and other diseases of the oral mucosa
* Insufficient prosthodontics
* Allergy against acrylic resin of prosthesis
* Allergy against Chinin-hydrochloride
* Xerostomia
* Pregnancy
* Psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2007-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Neurosensory differences between Burning Mouth Disorder patients and controls.
  The aim of the present study is to identify patients with idiopathic BMD. By way of qualitative and quantitative sensory testing (QST) and gustatory tests we want to find out whether neurosensory differences exist between patients with BMD and controls without any oral burning sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Peroz, PD Dr., Study Chair — Charité - Universitätsmedizin Berlin, Center for dental and craniofacial sciences, Department of restorative dentistry, Assmannshauser Str. 4-6, D-14197 Berlin; Markus R Fussnegger, Dr., Study Director — Charité - Universitätsmedizin Berlin, Center for dental and craniofacial sciences, Department of restorative dentistry, Assmannshauser Str. 4-6, D-14197 Berlin
Locations (1):
- Charité - Universitätsmedizin Berlin, Center for dental and craniofacial sciences, Department of restorative dentistry, Berlin, Germany

REFERENCES:
- [Background] Scala A, Checchi L, Montevecchi M, Marini I, Giamberardino MA. Update on burning mouth syndrome: overview and patient management. Crit Rev Oral Biol Med. 2003;14(4):275-91. doi: 10.1177/154411130301400405. PMID 12907696
- [Background] Forssell H, Jaaskelainen S, Tenovuo O, Hinkka S. Sensory dysfunction in burning mouth syndrome. Pain. 2002 Sep;99(1-2):41-7. doi: 10.1016/s0304-3959(02)00052-0. PMID 12237182
- [Background] Lauria G, Majorana A, Borgna M, Lombardi R, Penza P, Padovani A, Sapelli P. Trigeminal small-fiber sensory neuropathy causes burning mouth syndrome. Pain. 2005 Jun;115(3):332-337. doi: 10.1016/j.pain.2005.03.028. PMID 15911160
- [Background] Grushka M, Epstein JB, Gorsky M. Burning mouth syndrome and other oral sensory disorders: a unifying hypothesis. Pain Res Manag. 2003 Fall;8(3):133-5. doi: 10.1155/2003/654735. PMID 14657979
- [Background] Formaker BK, Frank ME. Taste function in patients with oral burning. Chem Senses. 2000 Oct;25(5):575-81. doi: 10.1093/chemse/25.5.575. PMID 11015329
- [Background] Bartoshuk LM, Snyder DJ, Grushka M, Berger AM, Duffy VB, Kveton JF. Taste damage: previously unsuspected consequences. Chem Senses. 2005 Jan;30 Suppl 1:i218-9. doi: 10.1093/chemse/bjh192. No abstract available. PMID 15738123